CLINICAL TRIAL: NCT05196152
Title: MomMoodBooster Randomized Components Trial: A Program for Perinatal Depressed Female Veterans
Brief Title: MomMoodBooster VA Program
Acronym: Perinatal MMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily Thomas, Clinical Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202102537; 202104724 (Other: HawkIRB)
Record Dates: First submitted 2021-11-19; First posted 2022-01-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Perinatal Depression; Postpartum Depression
Keywords: Postpartum Depression; Perinatal Depression; Veteran; Womens Mental Health
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either: 1) MomMoodBooster or 2) MomMoodBooster + phone coaching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MomMoodBooster Online (Active Comparator)
  Interventions: Behavioral: MomMoodBooster
- MomMoodBooster + Coach (Experimental)
  Interventions: Behavioral: MomMoodBooster; Behavioral: Phone Coaching

INTERVENTIONS:
Behavioral: MomMoodBooster — MomMoodBooster is an empirically validated online intervention for perinatal women.
Behavioral: Phone Coaching — Phone coaching calls occur weekly in conjunction with MomMoodBooster online modules.
  Arms: MomMoodBooster + Coach

SUMMARY:
The MomMoodBooster intervention is an empirically validated treatment for postpartum depression symptoms. The intervention was created by Brian Danaher and Milagra Tyler, who have continued to update the intervention technology and content. The intervention is now available for pregnant and postpartum Veterans, and it is accessible on browsers via computer, tablet, or mobile phone. The intervention contains six cognitive-behavioral modules that span six weeks, and it includes identification of pleasant activities, tracking mood and thoughts, and identification of goals. The current trial is an expansion of a nationwide service delivery project that has been ongoing for six years with the goal of offering the intervention to postpartum Veterans nationwide. Within that study, Veterans completed the online modules in concert with weekly phone coaching calls wherein coaches applied the content to the Veteran's current life. In addition, two booster modules and associated coaching calls were developed to continue application of the skills beyond the six-week intervention period. The present study seeks to investigate the incremental utility of the phone coaching component of the intervention by randomizing pregnant and postpartum Veterans to the MomMoodBooster intervention or the MomMoodBooster intervention plus phone coaching. Primary outcomes will include depressive symptoms, behavioral activation, and negative automatic thoughts.

DETAILED DESCRIPTION:
The purpose of the current study is to: 1) expand the MomMoodBooster intervention to pregnant Veterans and 2) to randomize Veterans to one of two intervention conditions. Veterans may be randomized to either 1) MomMoodBooster online intervention only or 2) MomMoodBooster online intervention and phone coaching. The study will examine the incremental utility of the phone coaching component of the intervention with the ultimate goal of VA-wide implementation. Veterans who report a history of or current mania or psychosis will be referred to mental health care locally. Patients who report elevated suicide risk will be directed to go to the nearest emergency room.

The study will recruit Veterans from around the nation. Investigators expect that 20% of female Veterans may be eligible. Based on national data, approximately 152,046 female Veterans in the USA are likely to have received care at a VA facility and are within the eligible age range. Centers for Disease Control and Prevention (CDC) data indicate that birth rates per 1000 women is 12.7. As such, about 3,866 female Veterans may be eligible per year. Veterans are eligible throughout the duration of pregnancy and up to 26 weeks postpartum.

Use of the medical record has proved successful in screening and enrolling postpartum Veterans nationwide. Veterans who are noted to be pregnant or postpartum in the VA medical record will be contacted to determine interest and eligibility.

Data will be obtained from the Veterans Health Administration (VHA) Corporate Data Warehouse through the VA Informatics and Computing Infrastructure, which includes pregnancy and postpartum diagnoses by the International Classification of Disease Tenth Revision Clinical Modification (ICD-9 and ICD-10 CM) codes, VHA outpatient visit dates, community care consults and medical services, patient demographics (such as race, ethnicity, date of birth, patient mailing address, and Rural-Urban Commuting Area Codes), and contact information. These data will be stored in a Microsoft Access database on VA servers, and the database will only be accessible to select members of the research team. The data will be imported to Access by a VA employee who does not have access to any participant data following enrollment. Demographic data are expected to be complete due to data being extracted from electronic medical records. All obstetric information will be verified in the screening process to ensure updated information is considered. Oversampling for rural Veterans will be conducted with the hopes of enrolling more rural Veterans (2:1 rural:non-rural Veteran ratio).

Veterans may also be referred through Maternity Care Coordinators (MCCs) or providers at VA medical centers. The MCCs may provide Veterans with the study's contact information or call the study team directly with the Veteran's permission. Veterans may also self-refer to the program by calling the research team or expressing interest via the MomMoodBooster website through the Contact link.

Based on VA medical records that identify a Veteran as being pregnant, Veterans will be mailed a letter detailing the study, and a return letter with prepaid envelope will be provided if the Veteran wishes to decline or express interest. If interest is expressed or if no return letter is received, a member of the research team will follow-up with a phone call to determine interest and answer questions. The study team will wait at least 5 days before following up with a phone call to ensure that the participant received the letter. The study team will call no more than 10 times without a returned phone call. A phone number is included in the letter so that Veterans can call and indicate that the Veteran is not interested in participating. The research team member will tell them about the study prior to screening if the Veteran is interested in being screened.

If interested, Veterans will be screened by phone. First, the study procedures will be reviewed orally. If a Veteran wishes to review the consent document prior to screening, the study team will mail her a copy of the consent form and call her 7 days later to review any questions and screen her if she remains interested. Veterans will be told that participation is entirely a personal choice, and participation has no bearing on healthcare at the VA or elsewhere. If a Veteran is not eligible at first screening, at the Veteran's request, the research team can call her in the future to re-screen, provided that the factor determining ineligibility is dynamic.

The screening will include access to internet/smartphone, less than 50 years of age, the PHQ-9 for depressive symptoms, basic demographic information, contact information, and the M.I.N.I. depression, mania, and psychosis modules. If a Veteran meets criteria (10 or more on the PHQ-9, no history or current mania, no history or current psychosis), a research team member will review the consent document and study procedures with her by phone. If she remains interested, a consent cover letter, consent document (one to sign and one for the Veteran's records), VA form for authorization to audio tape, VA HIPAA form, sociodemographic form, and baseline questionnaires will be mailed to her. Veterans will have until 26 weeks postpartum to consider whether the potential participant want to participate, at the end of which the person will no longer be eligible. Subjects will sign the VA 10-0493 HIPAA authorization form to give permission for access to medical records. Upon receipt of the signed forms and baseline questionnaires, forms will be reviewed by the research team. After completing the baseline assessment, the Veteran will be randomly assigned to condition -- either MMB online only or MMB + phone coaching. Veterans will then be assigned a phone coach. If a Veteran is assigned to MMB online only, the phone coach will call the Veteran for symptom monitoring during weeks 1, 3, and 5 of the intervention and administer the PHQ-9 by phone. If assigned to the phone coaching condition, the phone will call for all six weeks of the program to discuss the online content, and the PHQ-9 will be administered during weeks 1, 3, and 5 as well. Only members of the research team have access to study data, and files have restricted access to only the team members who require access.

The baseline questionnaire includes background and demographic information, the PHQ-9, the IDAS-II for internalizing symptoms, the BADS for behavioral avoidance and activation in depression, the Automatic Thoughts Questionnaire (ATQ) for negative automatic thoughts, the DAS for an individual's perception of the partner relationship, the Childhood Trauma Questionnaire (CTQ) for childhood trauma history, and a screening for military sexual trauma.

The program will be completed in 6-8 weeks. The program tracks use of the program, and this information is necessary for phone coaches to know whether a Veteran has logged in and completed relevant modules. This assists in the personalization of phone coaching calls.

After completion of the program, Veterans are offered the opportunity to complete two booster session modules at 14- and 20-weeks after enrollment. Participants in the MMB + phone coaching condition will receive two additional calls to discuss the booster session content, and Veterans who are in the online intervention only condition will receive two calls to monitor symptoms with the PHQ-9.

At any point in the program, if a Veteran expresses suicidality on the PHQ-9, the Columbia Suicide Severity Risk Scale will be administered by a member of the research team to determine suicide risk. If a Veteran is at high risk, the Veteran will be referred to emergency care. If the Veteran is not at high risk, recommendations will be developed with the Veteran to keep them safe and encourage connection with local providers.

Phone coaches are trainees who receive training and ongoing supervision in the intervention, interviewing, women's mental health, and the research protocol. The maximum number of calls per Veteran is 6 during the MMB portion of the intervention and 2 booster calls following completion of MMB. Duration of the calls is approximately 15-20 minutes. Reminders will be sent via text message about 24 hours prior to the scheduled call. Text messages will contain reminder of an appointment on [date] at [time] as well as the study phone number for reference if she has questions. Reminders to log into the program may occur via MyHealthEVet or by phone call. Calls will be audio recorded and saved on the University's secure data drive. The calls will be accessible by the research team. Recorded calls will be used for supervisory and training purposes, as well as coding of fidelity and competency.

After completion of the intervention, a follow-up survey will be mailed to the Veteran for completion at 3- and 6-months following enrollment. The follow-up questionnaires include PHQ-9, IDAS, BADS, ATQ, PSOC, DAS-8, and the Program Evaluation Questionnaire. If a Veteran prefers, the questionnaires can be completed by phone with a research team member. All interviews or coaching calls will be audiotaped to ensure fidelity. Veterans who report depressive symptoms in the mild or higher range (10 or more on PHQ-9) at follow-up will be referred to closest local VA for services.

Statistical analyses will compare differences between conditions over time using longitudinal modeling. The model will include condition (MMB, MMB + phone coach). Randomization will be stratified by pregnancy status (pregnant, postpartum).

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or within 26 weeks postpartum
* 18 - 50 years of age
* Experiencing elevated depressive symptoms at screening (PHQ-9 score of 10 or more)
* Have access to internet or smartphone

Exclusion Criteria:

* Past or current mania
* Current hypomania
* Past or current psychoses
* Active suicidality

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | Through study completion, an average of 6 months
  Symptoms of dysphoria, anhedonia, avolition, suicidality, lassitude, and changes in sleep and appetite are measured. The measure being utilized is the Inventory of Depression and Anxiety Symptoms, version 2 (IDAS-II). The 99 items are rated on a 5-point Likert scale from Not At All to Extremely. The measure of depressive symptoms used for this outcome is a 20-item composite, General Depression, and higher scores represent higher levels of depressive symptoms. Scores range from 20-100.
Change in Behavioral Activation | Through study completion, an average of 6 months
  The Behavioral Activation for Depression Scale, short form (BADS), assesses engagement with valued life domains. The scale has four subscales, including activation, avoidance/rumination, work/school impairment, and social impairment. The 25 items are rated on a 0-6 Likert scale, and items from the avoidance, work/school, and social subscales are reverse-scored. Total scores range from 0-150, with higher scores indicating higher engagement with personal values.
Change in Negative Automatic Thoughts | Through study completion, an average of 6 months
  This measure assesses the frequency of negative automatic thoughts. The 15 items are rated on a 1-4 Likert scale. Total scores range from 15-60, with higher scores indicating more frequent negative automatic thoughts.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms | Through study completion, an average of 6 months
  Symptoms of social anxiety, panic, traumatic intrusions, and traumatic avoidance are also measured with the Inventory of Depression and Anxiety Symptoms, version 2 (IDAS-II). The 99 items of this scale are rated on a 5-point Likert scale from Not At All to Extremely. The items are totaled to produce subscale scores with higher scores indicating higher levels of symptoms: Panic (8-40), Social Anxiety (6-30), Traumatic Intrusions (4-20), Traumatic Avoidance (4-20).
Change in Dyadic Adjustment | Through study completion, an average of 6 months
  The Dyadic Adjustment Scale (DAS) assesses satisfaction and support in the partner relationship, if the participant has a partner. The investigators are utilizing the Satisfaction subscale of the DAS. 7 items are rated on a 0-5 Likert scale, and the final item is rated on a 0-6 Likert scale. The total score ranges from 0 - 36, with higher scores indicating greater adjustment and satisfaction in the partner relationship.

OTHER OUTCOMES:
Program satisfaction | 6 months
  The program satisfaction questionnaire was developed to assess usability, confidence, and helpfulness that participants experienced with the MomMoodBooster program. Participants rate these items on a Likert scale, and qualitative feedback is also elicited. As this is a scale developed for program evaluation only, the scale is not meant to create a total score (i.e., individual items will be used as is.

CONTACTS AND LOCATIONS:
Overall Officials: Emily BK Thomas, PhD, Principal Investigator — University of Iowa; Rural Health Resource Center - Iowa City
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danaher BG, Milgrom J, Seeley JR, Stuart S, Schembri C, Tyler MS, Ericksen J, Lester W, Gemmill AW, Kosty DB, Lewinsohn P. MomMoodBooster web-based intervention for postpartum depression: feasibility trial results. J Med Internet Res. 2013 Nov 4;15(11):e242. doi: 10.2196/jmir.2876. PMID 24191345
- [Background] Kroska EB, Stowe ZN. Postpartum Depression: Identification and Treatment in the Clinic Setting. Obstet Gynecol Clin North Am. 2020 Sep;47(3):409-419. doi: 10.1016/j.ogc.2020.05.001. PMID 32762926
- [Background] Watson D, O'Hara MW, Naragon-Gainey K, Koffel E, Chmielewski M, Kotov R, Stasik SM, Ruggero CJ. Development and validation of new anxiety and bipolar symptom scales for an expanded version of the IDAS (the IDAS-II). Assessment. 2012 Dec;19(4):399-420. doi: 10.1177/1073191112449857. Epub 2012 Jul 20. PMID 22822173
- [Background] Fuhr K, Hautzinger M, Krisch K, Berking M, Ebert DD. Validation of the Behavioral Activation for Depression Scale (BADS)-Psychometric properties of the long and short form. Compr Psychiatry. 2016 Apr;66:209-18. doi: 10.1016/j.comppsych.2016.02.004. Epub 2016 Feb 9. PMID 26995255
- [Background] Solness CL, Kroska EB, Holdefer PJ, O'Hara MW. Treating postpartum depression in rural veterans using internet delivered CBT: program evaluation of MomMoodBooster. J Behav Med. 2021 Aug;44(4):454-466. doi: 10.1007/s10865-020-00188-5. Epub 2020 Oct 14. PMID 33052526
- [Background] Danaher BG, Milgrom J, Seeley JR, Stuart S, Schembri C, Tyler MS, Ericksen J, Lester W, Gemmill AW, Lewinsohn P. Web-Based Intervention for Postpartum Depression: Formative Research and Design of the MomMoodBooster Program. JMIR Res Protoc. 2012 Nov 22;1(2):e18. doi: 10.2196/resprot.2329. PMID 23612274
- [Background] Netemeyer, R. G., Williamson, D. A., Burton, S., Biswas, D., Jindal, S., Landreth, S., et al. (2002). Psychometric properties of shortened versions of the Automatic Thoughts Questionnaire. Educational and Psychological Measurement, 62, 111-129. https://doi.org/10.1177/0013164402062001008
- See also: MomMoodBooster — https://mommoodbooster.com/

DOCUMENTS (1):
  • Informed Consent Form (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT05196152/ICF_000.pdf